CLINICAL TRIAL: NCT03381859
Title: A Single-site, Open-label, Non-comparator Clinical Trial to eLiminate HCV-infection in Treatment-naïve, EgyptiAn Patients With End-stage Renal Disease on Renal Dialysis, With Chronic Hepatitis C Genotype 4 Infection Using a 12-week Course of Once-daily Single Oral Tablet of Elbasvir (50mg)/Grazoprevir (100 mg)
Brief Title: Clinical Trial to eLiminate HCV-infection in Treatment-naïve, Renally Impaired EgyptiAn Patients on Renal Dialysis, With Chronic Hepatitis C Genotype 4
Acronym: CLEAR-C4
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: HCV treatment expansion occurred in Egypt
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Cairo University (Other)
Responsible Party: Principal Investigator, Shyamasundaran Kottilil, Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00076974
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of
Keywords: Hepatitis C Virus; Genotype 4; End Stage Renal Disease
MeSH Terms: conditions — Hepatitis C; Kidney Failure, Chronic | interventions — elbasvir; grazoprevir; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Patients to receive 12 weeks of Elbasvir (50mg) / Grazoprevir (100mg)
  Interventions: Drug: Elbasvir/Grazoprevir 50 MG-100 MG Oral Tablet [ZEPATIER]

INTERVENTIONS:
Drug: Elbasvir/Grazoprevir 50 MG-100 MG Oral Tablet [ZEPATIER] — Hepatitis C Virus direct-acting antiviral

SUMMARY:
Primary Efficacy Objective

-To assess whether a 12-week treatment course with oral 50 mg elbasvir plus 100 mg grazoprevir given in a single daily dose to treatment-naïve patients with end-stage renal disease (ESRD) and infected with genotype 4 (GT4) chronic HCV (CHC) infection can produce a sustained viral response (SVR), i.e. HCV RNA below the lower limit of quantification [LLOQ] for 12 weeks (SVR12) after completion of the study treatment course

Secondary Objectives

* To assess the efficacy of elbasvir/grazoprevir in suppressing HCV viremia in treatment-naïve GT4 CHC patients at each scheduled visit and clinically meaningful endpoints (Week 2, 8 and 12 [End of Treatment - EOT]) and 24 (SVR12)
* To assess the safety and tolerability of a 12-week treatment course with elbasvir/grazoprevir in treatment-naïve patients with ESRD and infected with GT4 CHC.
* To assess liver fibrosis by non-invasive evaluation of liver stiffness (Fibroscan®) in the same patients before treatment and EOT and SVR12

Clinical hypotheses.

Primary Efficacy Hypothesis

- A 12-week treatment course with elbasvir/grazoprevir in treatment-naïve patients with ESRD and infected with GT4 CHC infection will result in an HCV RNA below the LLOQ in 95% of patients within 2 weeks of treatment, and at least 95% will have an SVR12.

Secondary hypotheses

* A 12-week treatment course with elbasvir/grazoprevir in ESRD GT4 treatment-naïve patients will result in undetectable viremia in 95% patients at Week 2, 4, 8 and 12 (EOT) and 24 (SVR12)
* Treatment will be safe and well-tolerated in these patients, as determined by the type and number of adverse events identified through laboratory testing, vital signs and physical examinations.
* In these patients with liver fibrosis before treatment, the liver fibrosis as assessed by non-invasive evaluation of liver stiffness (Fibroscan®) will improve by EOT and SVR12

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before undergoing any trial-related procedures
2. Male and female patients; age between 21 and 70 years inclusive
3. Chronic hepatitis C infection with genotype 4 confirmed by genotypic testing at screening or within 6 months of screening period
4. Treatment naïve - absence of prior failed treatment for HCV with Interferon plus ribavirin therapy or directly acting antivirals (treatment experienced)
5. Detectable HCV viral load (quantitative)
6. Liver cirrhosis subjects may be included but will be limited to those with compensated liver disease
7. Chronic kidney disease with end-stage liver disease (defined as glomerular filtration rate [eGFR] <=15 mL/min/1.73m2) on hemodialysis for at least 3 months, including individuals awaiting kidney transplant and those with failed kidney transplants but no longer on immunosuppressant therapy)
8. Screening laboratory values within the defined protocol thresholds
9. Women of child-bearing potential, must agree to abstinence or use of effective contraceptive methods (e.g. oral or injectable contraceptives, intra-uterine device (IUD), transdermal contraceptive patch) at least 2 weeks prior Day 1 through 14 days after the last dose of the study drug.
10. Ability to communicate, participate, and comply with the requirements of the entire study

Exclusion Criteria:

1. Patients didn't sign informed consent or under age of legal consent
2. Pregnant or breastfeeding woman
3. Has HCV genotypes other than G4
4. On peritoneal dialysis for management of kidney disease
5. Co-Infection with HIV and/or HBV (with positive HBsAg)
6. Evidence of hepatocellular carcinoma (HCC)
7. Evidence of hepatic decompensation as evidenced by presence or history of ascites, esophaegal or gastric bleeding, hepatic encelopathy or other signs of or symptoms of advanced liver disease, or cirrhotic subjects with Child-Pugh B or C, or who have a Purgh-Turcotte (CPT) score >6
8. Active or suspected non-hepatic malignancy or history of any malignancy except for cured basal cell or squamous cell skin cancer or in situ cervical cancer
9. Organ transplant (including hematopoietic stem cell transplant) other than kidney, cornea, and hair
10. Conditions requiring, or likely to require, chronic systemic administration of corticosteroids during the course of the trial
11. Uncontrolled or poorly controlled hypertension
12. Pregnant, breast-feeding, expecting to conceive or donate eggs, or donate sperm from Day 1 through 14 days after the last study dose.
13. Significant cardiovascular disorder (e.g. myocardial infarction or unstable angina) or interventional cardiovascular procedure within 3 months prior to signing informed consent
14. Recent (within 3 months prior to signing informed consent) episode or recurrence of stroke, transient ischemic attack (TIA) or neurological disorder, including but not limited to seizures
15. ALT or AST > 10-fold the upper limit of normal
16. Evidence of liver disease due to causes other than chronic HCV infection
17. Evidence of poorly controlled diabetes (defined as HbA1c > 8%)
18. History of alcohol or drug abuse within the last 12 months
19. Serum albumin level < 3.0 g/dL
20. INR > 1.3 N
21. Total Bilirubin levels > 2.0 mg/dL unless explained by Gilbert's disease
22. Platelets Count <75,000/µL
23. White blood cell count < 1500 µL (mm3)
24. Clinically significant TSH and T4 level poorly controlled thyroid function
25. Patients with any abnormality on physical examination, vital signs (sitting systolic blood pressure greater than 150 mmHg, sitting diastolic blood pressure greater than 90 mmHg and pulse greater than 90 bpm) and ECG, unless these abnormalities are judged to be not clinically significant by the Investigator
26. Body Mass Index < 18.5 or > 35 kg/m2
27. Use of other investigational drugs/treatments within the previous 3 months
28. Known hypersensitivity to any of the test materials or related compounds.
29. Active autoimmune disease.
30. History of moderate, severe or uncontrolled psychiatric disease, especially severe depression and prior suicidal attempt.
31. Unable to comply with research study visits.
32. Poor venous access not allowing screening laboratory collection.
33. Any other condition that, in the opinion of the Investigator, may be a contraindication to study participation or jeopardize the study conduct according to the protocol.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
SVR12 | 24 weeks from treatment initiation date
  absence of HCV plasma RNA 12 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shyamasundaran Kottilil, MD, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Kasr Alainy Hospital, Cairo, Almanial, Egypt

IPD SHARING:
Plan to Share IPD: No